CLINICAL TRIAL: NCT02267798
Title: The Effects of Repetitive Arm Training Combined With Functional Electrical Stimulation on Upper Extremity Motor Recovery in Sub-acute Stroke Survivors
Brief Title: Repetitive Arm Training + FES on Upper Extremity Motor Recovery in Sub-acute Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, MD, MD, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Regionale WP1
Record Dates: First submitted 2014-01-16; First posted 2014-10-20 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Stroke; Arm Motor Recovery
Keywords: Stroke; Rehabilitation; Arm motor recovery; biological biomarkers
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- arm training combined with FES (Experimental): Arm training protocol Training sessions will last for 60 minutes and will focus on repetitive tasks that incorporate multidirectional reaching actions. In this robot-assisted therapy a robot manipulator applies forces to the paretic arm during goal-directed movements.
  Functional electrical stimulation protocol Experimental group will receive up to 40 minutes of FES after arm training. The device consists of a battery powered programmable stimulator and a forearm-wrist-hand orthosis containing 5 electrodes positioned to provide reliable activation of muscles. The intensity of stimulation will be set to a level that provided comfortable and consistent activation of the extensor and flexor muscles to achieve whole hand opening and functional grasping.
  Interventions: Device: arm training combined with FES
- conventional therapy (Active Comparator): The conventional rehabilitation program will consist of physiotherapy sessions (100 min/day) following an individualized approach. The program aims at the restoration of mobility and daily living competence, Specific exercises for the affected upper limb will include, bilateral tasks and facilitation techniques based on neuro-developmental treatment.
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: conventional therapy — The conventional rehabilitation program will consist of physiotherapy sessions (100 min/day) following an individualized approach. The program aims at the restoration of mobility and daily living competence. Specific exercises for the affected upper limb will include, bilateral tasks and facilitation techniques.
  The amount of treatment will to be comparable between control and experimental groups in order to avoid possible confounding factors.
  Arms: conventional therapy
Device: arm training combined with FES — Arm training protocol Training sessions will last for 60 minutes. The Reo Therapy System is robot-assisted therapy; during the session the subject's affected hand is placed on or strapped onto a robotic arm and the subject is instructed to either actively reach predefined reach points, or to be guided while the robotic arm leads the arm towards these reach points.
  Functional electrical stimulation protocol Experimental group will receive up to 40 minutes of FES after arm training. The device consists is a stimulator containing 5 electrodes positioned to provide reliable activation of the following muscles: extensor digitatum communis and extensor pollices brevis, flexor pollices longus, flexor digitatum superficialis, and thenar muscles.
  Arms: arm training combined with FES

SUMMARY:
Rehabilitation restores functions and reduces disabilities due to diseases sequelae. The relationship between intensity of rehabilitation and clinical outcomes, recently emphasized, has generated a great interest for technological high-intensity interventions. However, their effects compared to traditional interventions as well the involved biological mechanisms remain uncertain. The present Strategic Program aims to predict the treatment efficacy in specific rehabilitation profiles, to improve the use of "targeted" therapies and the individual management of patients affected by stroke and to transfer these findings into rehabilitative strategies.

DETAILED DESCRIPTION:
Primary endpoint: Fugl-Meyer Upper Extremity (FM-UE) Secondary endpoints: Box and Block Test (BBT), Modified Ashworth Scale (MAS); motor cortex excitability (TMS); Electromyography analysis of muscle activation patterns during upper extremity movements; measurements of cerebral perfusion (NIRS); circulating biomarkers (see Figure 3 and Table 1). Overall assessments will be performed pre-, mid-, post-treatment and at 6-months follow-up.

ELIGIBILITY:
Inclusion criteria:

* males and females, age 18 to 79 years
* diagnosis of first, single unilateral ischemic stroke verified by brain imaging < 8 weeks
* upper limb motor function defined by an FM-UE score > 11 and <55

Exclusion criteria:

* medical conditions likely to interfere with the ability to safely complete the study protocol
* impaired cognitive functioning: score less than 24 on the Mini Mental Status Examination (MMSE)
* severe upper-limb pain, referred as > 7 at Visual Analog Scale (VAS)
* history of seizures or epilepsy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Fugl-Meyer Upper Extremity (FM-UE) | 1) One week prior to treatment initiation 2) after 3 weeks 3) the week after the end of treatment 4) at 6 months follow-up.
  Measure of upper extremity motor impairment. The upper extremity score ranges from 0-66.

SECONDARY OUTCOMES:
Wolf Motor Function Test (WMFT) Manual | 1) One week prior to treatment initiation 2) after 3 weeks 3) the week after the end of treatment 4) at 6 months follow-up
Modified Ashworth Scale (MAS)for spasticity measure | 1) One week prior to treatment initiation 2) after 3 weeks 3) the week after the end of treatment 4) at 6 months follow-up
  MAS: a 6-point measure of spasticity. We will assess the spasticity at the shoulder, elbow and, wrist
Motor Activity Log (MAL)measures change in arm use during activities of daily living | 1) One week prior to treatment initiation 2) after 3 weeks 3) the week after the end of treatment 4) at 6 months follow-up
  Motor Activity Log (MAL): assessment of the change in real-world arm use in activities of daily living. Subjects are asked to score the quality of movement as well as amount of use of the affected arm in a number of common daily activities
Functional Independence Measure (FIM) | 1) One week prior to treatment initiation 2) after 3 weeks 3) the week after the end of treatment 4) at 6 months follow-up
  FIM measures level of independence during activities of daily living.
Stroke Impact Scale 3.0 (SIS) | 1) One week prior to treatment initiation 2) after 3 weeks 3) the week after the end of treatment 4) at 6 months follow-up
  Assesses health status following stroke
Box and Block test | 1) One week prior to treatment initiation 2) after 3 weeks 3) the week after the end of treatment 4) at 6 months follow-up
  It counts the number of blocks that can be transported from one compartment of a box to another compartment within 1 min.
Motor cortex excitability (single pulse and paired pulse TMS) | 1) One week prior to treatment initiation 2) after 3 weeks 3) the week after the end of treatment 4) at 6 months follow-up
  1. Single pulse TMS Single-Pulse TMS will be used to study cortical-spinal tract excitability in primary motor cortex (M1).
  2. Paired-pulse TMS Paired-Pulse TMS will be used to study intracortical excitability.
Analysis of muscle activation patterns during upper extremity movements | 1) One week prior to treatment initiation 2) the week after the end of treatment 3) at 6 months follow-up
  A measure of the coordination of muscular activity across muscles of the upper limbs will be derived from recordings performed during a series of upper extremity motor tasks.
NIRS (Near Infrared Spectroscopy) | 1) One week prior to treatment initiation 2) after 3 weeks 3) the week after the end of treatment 4) at 6 months follow-up
  For the NIRS it will use an 32-channel NIRS imaging equipment which consist of 16 pairs of emitting and detecting optical fibers attached to a custom-made head cap placed on primary motor cortex.
  NIRS measurements will be performed during 6 cycles of 15s hand reaching and grasping and 45s resting while sitting on a chair.
Circulating Biomarkers | 1) One week prior to treatment initiation 2) after 3 weeks 3) the week after the end of treatment 4) at 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nino Basaglia, MD, Principal Investigator — Ferrara University Hospital
Locations (2):
- Italy (2):
  - Physical Medicine and Rehabilitation Department Ferrara, Ferrara, Emilia-Romagna
  - Ferrara University Hospital, Ferrara, Ferrara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Straudi S, Baroni A, Mele S, Craighero L, Manfredini F, Lamberti N, Maietti E, Basaglia N. Effects of a Robot-Assisted Arm Training Plus Hand Functional Electrical Stimulation on Recovery After Stroke: A Randomized Clinical Trial. Arch Phys Med Rehabil. 2020 Feb;101(2):309-316. doi: 10.1016/j.apmr.2019.09.016. Epub 2019 Nov 1. PMID 31678222